CLINICAL TRIAL: NCT03438097
Title: Survey of Non-resuscitation Fluids in Septic Shock
Acronym: SURF
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, peter bentzer, Associate professor, Region Skane
Other Study IDs: ICU Skane 2017
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Septic Shock
Keywords: Fluid therapy; Non-resuscitation fluids; Septic shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to survey the type and the amount of non-resuscitation fluids that patients with septic shock receives during their first 5 days of ICU admission.

DETAILED DESCRIPTION:
Background: Several studies indicate that a large part of the fluid intake in intensive care patients consists of fluids that are given for indications other than volume expansion. However, the type of non-resuscitation fluids that hemodynamically unstable ICU patients receive has not been well characterized.

Methods: A multicenter observational cohort study. Baseline data including, sex, age, physiological data at admission, source of sepsis, illness severity, and ICU and hospital mortality will be collected.

Fluids administered during the first five days of ICU admission will be registered. Fluids used as vehicle to administer drugs will be regarded as non-resuscitation fluids and will be characterized in detail. All glucose solutions will be regarded as non-resuscitation fluids. Crystalloids delivered at a rate of < 5 ml/kg/h will be considered as non-resuscitation fluids. Parenteral nutrition will be regarded as non-resuscitation fluids. Crystalloids delivered at a rate of ≥ 5 ml/kg/h will be considered to be resuscitation fluids. Blood products and colloids will be regarded as resuscitation fluids.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock per SEPSIS-3 criteria within 24 hrs of ICU admission
* Informed consent from patient or next of kin if required by local ethical review Board

Exclusion Criteria:

• Lack of informed consent (see above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted with septic shock during a 4 month period in ICUs in Sweden and in British Columbia, Canada. A maximum of 30 patients per centre will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Type, indication and volume of fluids given to septic shock patients for other reasons than circulatory support. | First five days in ICU
  Type of fluid is defined as either 0.9% normal saline, glucose, Ringers acetate/lactate, enteral nutrition, parenteral nutrition or sterile water.
  Indication is defined as vehicle, nutrition, maintenance or other. Volume will be reported in ml.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, MD, PhD, Principal Investigator — Lund University, Lund, Sweden
Locations (9):
- Canada (2):
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
- Sweden (7):
  - ICU Halmstad Hospital, Halmstad
  - ICU Helsingborg Hospital, Helsingborg
  - ICU Kristianstad Hospital, Kristianstad
  - ICU Skane University Hospital, Lund
  - Department of Infections Diseases, Malmo
  - ICU Skane University Hospital, Malmo
  - ICU Ystad Hospital, Ystad

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol can be shared from March 1st. Clinical Study Report (CSR) can be shared as data analysis is complete.
Access Criteria: On reasonable request